CLINICAL TRIAL: NCT05995457
Title: Efficacy of the Combination of " Z-track " and " Airlock " Techniques During Intramuscular Injection of Haloperidol Decanoate in Adult Patients With Schizophrenic or Related Disorder : A Multicenter Randomized Controlled Trial
Brief Title: The IM-ZBULLE Study : " Z-track " and " Airlock " Techniques During Intramuscular Injection of Haloperidol Decanoate
Acronym: IM-ZBULLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Groupe Hospitalier Paul Guiraud (Unknown); Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D23-P001
Record Dates: First submitted 2023-07-18; First posted 2023-08-16 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia; Psychosis
Keywords: Schizophrenia; Haloperidol decanoate
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Advanced practice nurses (APNs) will carry out clinical examinations before and after the treatment. They will not be present during the treatment, and the patient will not know the technique used, in order to ensure a double-blind evaluation. Only the nurses performing the injection will be aware of the technique used (experimental or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramuscular injection of Haloperidol decanoate using the "Z-track" and "Airlock" techniques (Experimental): Intramuscular injection involves administering the drug treatment Haloperidol decanoate into muscle tissue using the "Z-track" and "Airlock" techniques.
  Interventions: Other: Intramuscular injection of Haloperidol decanoate using the "Z-track" and "Airlock" techniques
- Control arm, Intramuscular injection as usual (Other): Intramuscular injection involves administering the drug Haloperidol decanoate into muscle tissue using the usual technique
  Interventions: Other: Intramuscular injection of Haloperidol decanoate using standard techniques

INTERVENTIONS:
Other: Intramuscular injection of Haloperidol decanoate using the "Z-track" and "Airlock" techniques — Intramuscular injection involves administering the drug treatment Haloperidol decanoate into muscle tissue using the "Z-track" and "Airlock" techniques
  Arms: Intramuscular injection of Haloperidol decanoate using the "Z-track" and "Airlock" techniques
Other: Intramuscular injection of Haloperidol decanoate using standard techniques — Intramuscular injection involves administering the drug Haloperidol decanoate into muscle tissue using the usual technique.
  Arms: Control arm, Intramuscular injection as usual

SUMMARY:
Intramuscular injection (IMI) is the process of administering a drug treatment into muscle tissue. The transmission of skills in this care practice is essentially based on the experience of peers. In France, there are no official guidelines for this technical procedure.

Haloperidol decanoate is widely used in psychiatry. This long-acting antipsychotic treatment considerably reduces the risk of relapse and hospitalization. It is administered by IMI. This treatment is invasive, painful and risks complications for the patient. Nurses must ensure that the treatment is as painless as possible, and adapt their practice in line with current recommendations.

Among the various IMI techniques available, the "Z-track" and the "Airlock" limit leakage into subcutaneous tissues when the needle is withdrawn, by locking the active product into the muscular tissues. According to an exploratory study (n=303), 73% of nurses observe active product leakage after injections, and 89% of nurses are not familiar with either the "Z-track" or "Airlock" techniques.

Many foreign studies have been carried out to demonstrate the relevance of these techniques, particularly in terms of pain reduction during treatment, but the results have yet to be confirmed.

The investigators hypothesize that the combined use of the "Z-track" and "Airlock" techniques during intramuscular injection of Haloperidol decanoate is more effective in reducing patient pain than usual practice.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind, controlled, study in 2 parallel groups.

Experimental and control administration protocols will be standardized to harmonize injection practices between the different nurses providing care, and to control some variables. Nurses will have been trained in these protocols and in experimental injection techniques.

The experimental group will be offered an intramuscular injection using the "Z-track" and "Airlock" techniques, while the control group will have an "usual" injection.

An intermediate analysis of futility and efficacy is planned once 50% of the planned sample has completed the study.

The object of the research is the intramuscular injection procedure - Product injected: haloperidol decanoate (Haldol Decanoas®).

ELIGIBILITY:
Inclusion Criteria:

* Adult ;
* having an outpatient treatment in a Mental Health Community Center ("Centre Médico-Psychologique" CMP in french) ;
* with an CIM-10 diagnosis between F20-F29 (Schizophrenia, schizotypal disorder and delusional disorders);
* communicative and able to give free and informed consent to the study;
* prescribed Haloperidol decanoate;
* covered by the french social security

Exclusion Criteria:

* Minor ;
* pregnant women ;
* with insufficient understanding of the French language to understand the VAS;
* suffering from any of the following known somatic comorbidity : coagulation disorder, leucopenia, immunosuppression;
* currently prescribed treatment: immunosuppressant, anticoagulant, antibiotic, antiretroviral, other products administered by IMI at dorsogluteal injection sites (antibiotic therapy, hormone therapy, vitamin therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
pain reduction | Day 0 intervention day T
  To evaluate the efficacy of combining the "Z-track" and "Airlock" techniques concerning reducing pain in adult patients treated with Haloperidol decanoate. The primary outcome measure is pain reduction, assessed using a millimeter-scale visual analogic scale (VAS) to measure pain perceived by the patient 5 minutes after the treatment. The score is between 0 (minimum) and 10 (maximum) centimeters. The higher the score, the worse the result.

SECONDARY OUTCOMES:
Drug leakage reduction | Day 0 intervention day
  To measure the loss (leakage) of active product when the needle is withdrawn : The outcome measure is a reduction in the loss of active product by assessing the diameter (using a millimeter scale) of active product that flow back through the puncture site using an absorbent pad.
Impact of the injection | Day 0 to Day 3
  To measure the impact of combining the "Z-track" and "Airlock" techniques on potential complications related to treatment : The outcome measure is the reduction in signs of secondary complications, as measured by a pre- and post-injection clinical examination and a phone call to the patient between Day 1 and Day 3.
Improving participants satisfaction | Day 14 or Day 21 or Day 28 depending to the frequency established by the prescription1
  To measure overall patient satisfaction with the combination of "Z-track" and "Airlock" intramuscular injection techniques. The outcome measure is participant satisfaction, assessed using Attkisson's CSQ-8 questionnaire. This scale comprises 8 questions. Depending on the answer, each question awards 1 to 4 points. The score is therefore between 8 (minimum) and 32 (maximum) points. The higher the score, the better the result.
Improving the therapeutic alliance | Day 0 (intervention day) and Day 14 or Day 21 or Day 28 depending to the frequency established by the prescription
  To measure therapeutic alliance during follow-up :The outcome measure is the overall therapeutic alliance score, using the Working Alliance Inventory (WAI) scale before and after intervention. This scale comprises 12 questions. Each question awards 1 to 5 points, depending on the answer. The score is between 12 (minimum) and 60 (maximum) points. The higher the score, the better the result.
Identifying the obstacles and levers to changing practices | During 14 Months
  To identify the levers and obstacles to nurses' change of practice : The outcome measure is the identification of levers and obstacles to change in professional practice among psychiatric nurses, by means of a complementary qualitative descriptive study.

CONTACTS AND LOCATIONS:
Overall Officials: Rayan BCHINI, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (1):
- Rayan BCHINI, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bchini R, Goutte N. [Evidence-based practice and nursing: intramuscular injection in psychiatry]. Soins Psychiatr. 2023 May-Jun;44(346):21-26. doi: 10.1016/j.spsy.2023.04.006. Epub 2023 Jun 7. French. PMID 37328226
- [Background] Rodger MA, King L. Drawing up and administering intramuscular injections: a review of the literature. J Adv Nurs. 2000 Mar;31(3):574-82. doi: 10.1046/j.1365-2648.2000.01312.x. PMID 10718876
- [Background] Wynaden D, Landsborough I, Chapman R, McGowan S, Lapsley J, Finn M. Establishing best practice guidelines for administration of intra muscular injections in the adult: a systematic review of the literature. Contemp Nurse. 2005 Dec;20(2):267-77. doi: 10.5172/conu.20.2.267. PMID 16393108
- [Background] Sanlialp Zeyrek A, Takmak S, Kurban NK, Arslan S. Systematic review and meta-analysis: Physical-procedural interventions used to reduce pain during intramuscular injections in adults. J Adv Nurs. 2019 Dec;75(12):3346-3361. doi: 10.1111/jan.14183. Epub 2019 Sep 13. PMID 31452229
- [Background] Keen MF. Comparison of intramuscular injection techniques to reduce site discomfort and lesions. Nurs Res. 1986 Jul-Aug;35(4):207-10. PMID 3636818
- [Background] Kim KS. [Comparison of two intramuscular injection technics on the severity of discomfort and lesions at the injection site]. Kanho Hakhoe Chi. 1988 Dec;18(3):257-68. doi: 10.4040/jnas.1988.18.3.257. Korean. PMID 3230758
- [Background] Quartermaine S, Taylor R. A comparative study of depot injection techniques. Nurs Times. 1995 Jul 26-Aug 1;91(30):36-9. PMID 7644369
- [Background] Mac Gabhann L. A comparison of two depot injection techniques. Nurs Stand. 1998 Jun 3-9;12(37):39-41. doi: 10.7748/ns1998.06.12.37.39.c2512. PMID 9732632
- [Background] Yilmaz DK, Dikmen Y, Kokturk F, Dedeoglu Y. The effect of air-lock technique on pain at the site of intramuscular injection. Saudi Med J. 2016 Mar;37(3):304-8. doi: 10.15537/smj.2016.3.13113. PMID 26905354
- [Background] Kara D, Yapucu Gunes U. The effect on pain of three different methods of intramuscular injection: A randomized controlled trial. Int J Nurs Pract. 2016 Apr;22(2):152-9. doi: 10.1111/ijn.12358. Epub 2014 Jul 11. PMID 25039702
- [Background] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Background] Heshmatifar N, Salari M, Rad M, Afshari Saleh T, Borzoee F, Rastaghi S. A New Approach on the pain management of intramuscular injection: A Triple-Blind Randomized Clinical Trial. Pain Manag Nurs. 2022 Jun;23(3):353-358. doi: 10.1016/j.pmn.2021.01.010. Epub 2021 Mar 11. PMID 33714700
- [Background] Bloch Y, Mendlovic S, Strupinsky S, Altshuler A, Fennig S, Ratzoni G. Injections of depot antipsychotic medications in patients suffering from schizophrenia: do they hurt? J Clin Psychiatry. 2001 Nov;62(11):855-9. doi: 10.4088/jcp.v62n1104. PMID 11775044